CLINICAL TRIAL: NCT03793699
Title: Evaluation of the Links Between Sleep Disorders and the Risk of Suicide Attempt
Acronym: HYPNOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2017_55; 2017-A03649-44 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-10-16; First posted 2019-01-04 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Attempted Suicide
Keywords: Suicide; Suicidal ideation; Sleep disorder
MeSH Terms: conditions — Suicide, Attempted; Suicide; Suicidal Ideation; Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group : realized a suicide attempt: adults having realized a suicide attempt and without histories of suicide attempt.
- control group : only suicidal ideas: adults having suicidal ideas without suicidal acting out and without histories of suicide attempt.

SUMMARY:
Several studies have demonstrated an association between sleep disorders such as insomnia and nightmares to suicidal ideations and behaviors.

Nevertheless, some of these studies are methodologically questionable especially in the exploration of sleep disorders. Furthermore, confounding factors such as depressive symptomatology are not controlled and the measurement of suicidal behavior has often been taken into account as a historical measure, not as a current event, which introduces uncertainties and a lack of precision regarding the temporality of the phenomena.

Today, while the links between sleep disorders and suicidal risk are well known, we have a lack of information on the importance and the role of sleep disorders as a precipitating factor. Indeed, few studies have evaluated the temporal link between sleep disorders and suicidal acts.

The objective of this study is to evaluate the links between acute and chronic sleep disorders and the risk of suicide attempt

DETAILED DESCRIPTION:
Pilot, prospective, monocentric case-control study.

There are 2 groups of subjects :

* group of patients who have made a suicide attempt
* control group with only suicidal ideas

First visit V1 is performed within the first 72 hours of hospitalization. A re-assessment is scheduled 1 month after (V2).

At V1, collected parameters are : chronic sleep disorders, chronotype, specific sleep disorders in posttraumatic stress disorder, nightmares and the distress associated, childhood trauma, cognitive dysfunction, suicidal ideation and psychopathologic assessment.

At V2, we assess evolution of sleep disturbances and suicidal ideation.

ELIGIBILITY:
Inclusion Criteria

Criterion specific to the studying group :

- Subjects hospitalized and whose indication of hospitalization is a suicide attempt by voluntary drug intoxication or phlebotomy during the last 72 hours, without any history of attempted suicide

Criterion specific to the control group:

- Subjects hospitalized since less than 72 hours, and whose indication of hospitalization is the presence of suicidal ideas, without any history of attempted suicide

Exclusion Criteria:

* Pregnant of lactating women
* Diagnosed dementia pathology
* Proven intellectual disability
* Patient whose physical or mental state does not allow the passing of the tests of the study
* Under protective measures (guardianship/supervision)
* Refusal to participate in the study
* Diagnosed with chronic or severe psychiatric illness (psychotic disorder, bipolarity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population in the study is a population of adults having realized a suicide attempt and without histories of suicide attempt. She(it) will be compared with a population of adults having suicidal ideas without suicidal acting out and without histories of suicide attempt.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-02-04 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Sleep disorders intensity by the Insomnia Severity Index (ISI) | at the 48 hours after the hospitalization; at the maximum within 72 hours.
  ISI score in the last 2 weeks between a group of suicide attempts and a group with suicidal thoughts suicidal The Insomnia Severity Index has seven questions. The seven answers are added up to get a total score.

SECONDARY OUTCOMES:
Correlation between Beck Suicide Intent Scale (BSIS) score and ISI score | Baseline (visit inclusion) and at one month ago
  Correlation between Beck Suicide Intent Scale (BSIS) score and ISI score The Suicide Intent Scale (SIS) wconsists of 15 questions which are scaled from 0-2, which take into account both the logistics of the suicide attempt as well as the intent. The scale has high reliability and validity. Completed suicides ranked higher in the severity of the logistics than attempted suicides (it was impossible to measure intent for the completed suicides), and those with multiple attempts had higher scores than those who only attempted suicide once
Evolution of ISI score | At one month +/- 15 days ant at 3 months +/-3 weeks
  Assess the evolution of sleep disturbances for each group by ISI Score
Chronotype classification by MCTQ | at the 48 hours after the hospitalization; at the maximum within 72 hours;at 3 months +/-3 weeks
  Exploratory descriptive measures in the 2 groups
Pittsburg Sleep Quality Index (PSQI) score | at the 48 hours after the hospitalization; at the maximum within 72 hours,at 3 months +/-3 weeks
  PSQI score between the groups PSQI is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete.
Childhood Trauma Questionnaire (CTQ) score | at the 48 hours after the hospitalization; at the maximum within 72 hours.
  CTQ score between the groups The Childhood Trauma Questionnaire was developed as a screening tool for histories of abut and neglect. The self-report includes a 28-item test that measures 5 types of maltreatment - emotional, physical, and sexual abuse, and emotional and physical neglect.
Montréal Cognitive Assessment (MocA) | at the 48 hours after the hospitalization; at the maximum within 72 hours.
  cognitive assessment by Moca test

CONTACTS AND LOCATIONS:
Overall Officials: Vincent JARDON, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Fontan, CHU, Lille, France